CLINICAL TRIAL: NCT02951169
Title: Multicenter Cohort Study: To Explore the Standard Surgical Indication in Gallbladder Benign Disease
Brief Title: Exploration of Standard Surgical Indication in Gallbladder Benign Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Shen Kang Hospital Development Center (Other)
Responsible Party: Principal Investigator, Zhaohui Tang, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-034
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Gallbladder Stone; Cholecystitis; Gallbladder Polyps
MeSH Terms: conditions — Cholecystolithiasis; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — No intervention. Treatment are accordance with clinical practice.

SUMMARY:
This study evaluates life quality of patients who were diagnosed with gallbladder benign disease through Gastrointestinal Quality of Life Index (GIQLI) scale. Researchers will establish a database including 20,000 patients. Through observational followup and statistic analysis，identifing a model or scale to standardized surgical indication, help surgeons and patients determine the best treatment decision.

DETAILED DESCRIPTION:
The incidence of gallbladder benign diseases are increasing today. Most patients are accepting cholecystectomy. Is it better postoperation for this sort of patients? In other words, there is no specific indication for cholecystectomy in gallbladder benign diseases. Investigators want to explore the specific surgical indication for these patients so that surgeons could help patients make the best decision according to our evaluation model. This model may be a scale that summarizes and quantizes correlative factors of individual, which will be discussed by statisticians and experts of biliary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gallbladder benign disease, including gallbladder stone、cholecystitis and polypoid lesions of gallbladder from December 2016 to September 2018.
* Have been clearly informed the purpose of this study, methods and other information, voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

* Complicated with bile duct stones and other biliary tract disease or suspected with gallbladder carcinoma、biliary tract cancer.
* Complicated with severe diseases such as organ dysfunction that cannot accept surgery
* Abdominal operation history.
* Pregnant or lactation.
* Coagulopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed with Gallbladder Benign Disease.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Life Quality (Through GIQLI:Gastrointestinal Quality of Life Index) | Every three months, up to 18 months
  Patients with surgery must including preoperative score

SECONDARY OUTCOMES:
The Rate of Accidentally Gallbladder Carcinoma During Cholecystectomy | Through study completion, an average of 18 months
The Rate of Abdominal Pain After Cholecystectomy | Through study completion, an average of 18 months
The Rate of Diarrhea After Cholecystectomy | Through study completion, an average of 18 months
The Rate of Abdominal Distension After Cholecystectomy | Through study completion, an average of 18 months
Hospital Stay | Through study completion, an average of 18 months
Total Expense of Patients Including Medication、Operating Costs and Check-Up Expense | Through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Tang, Phd, MD, Principal Investigator — Xinhua Hospital,School of Medicine,Shanghai Jiao Tong University
Locations (1):
- Zhang Yong, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Database including 20000 patients diagnosed with gallbladder benign disease will be available in the website and investigators' article.

REFERENCES:
- [Result] da Costa DW, Bouwense SA, Schepers NJ, Besselink MG, van Santvoort HC, van Brunschot S, Bakker OJ, Bollen TL, Dejong CH, van Goor H, Boermeester MA, Bruno MJ, van Eijck CH, Timmer R, Weusten BL, Consten EC, Brink MA, Spanier BWM, Bilgen EJS, Nieuwenhuijs VB, Hofker HS, Rosman C, Voorburg AM, Bosscha K, van Duijvendijk P, Gerritsen JJ, Heisterkamp J, de Hingh IH, Witteman BJ, Kruyt PM, Scheepers JJ, Molenaar IQ, Schaapherder AF, Manusama ER, van der Waaij LA, van Unen J, Dijkgraaf MG, van Ramshorst B, Gooszen HG, Boerma D; Dutch Pancreatitis Study Group. Same-admission versus interval cholecystectomy for mild gallstone pancreatitis (PONCHO): a multicentre randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1261-1268. doi: 10.1016/S0140-6736(15)00274-3. PMID 26460661
- [Result] Shabanzadeh DM, Sorensen LT, Jorgensen T. A Prediction Rule for Risk Stratification of Incidentally Discovered Gallstones: Results From a Large Cohort Study. Gastroenterology. 2016 Jan;150(1):156-167.e1. doi: 10.1053/j.gastro.2015.09.002. Epub 2015 Sep 14. PMID 26375367
- [Result] Cotton PB, Durkalski V, Romagnuolo J, Pauls Q, Fogel E, Tarnasky P, Aliperti G, Freeman M, Kozarek R, Jamidar P, Wilcox M, Serrano J, Brawman-Mintzer O, Elta G, Mauldin P, Thornhill A, Hawes R, Wood-Williams A, Orrell K, Drossman D, Robuck P. Effect of endoscopic sphincterotomy for suspected sphincter of Oddi dysfunction on pain-related disability following cholecystectomy: the EPISOD randomized clinical trial. JAMA. 2014 May;311(20):2101-9. doi: 10.1001/jama.2014.5220. PMID 24867013